CLINICAL TRIAL: NCT04352712
Title: Growth Hormone Modulated Gene Expression in Monocytes of Healthy and Growth Hormone Deficient Children
Brief Title: Gene Expression in Monocytes of Growth Hormone Deficient Children
Acronym: GEMGH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Mario Vitale, Professor, University of Salerno
Other Study IDs: GHUSalerno
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Children: healthy children, untreated, donors of monocytes
  Interventions: Other: blood sampling
- GHD children: GHD children, untreated, donors of monocytes
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling

SUMMARY:
The Growth hormone (GH) is mainly synthesized in the anterior portion of the pituitary gland and has an effect on different body areas. Secreted in the circulatory stream, growth hormone reaches the liver and here stimulates the secretion of somatomedin C better known as insulin-like growth factor 1 (IGF), which constitutes its main anabolic effector.

Growth hormone deficiency (GHD) is characterized by a delay in the statural growth in children and is correlated with a worsening of body composition, cognitive functions, lipid metabolism, bone mineralization, cardiac performance and exercise in adults. Recombinant GH (rhGH) replacement therapy can correct these alterations and therefore improve the quality of life in treated patients, and accelerate growth in children.

The optimal dosage of rhGH varies for each patient, as the response to treatment suffers from considerable inter-individual variability. To date, IGF1 is the only available biomarker whose plasma levels correlate with replacement therapy.

It is important to underline how somatomedin C does not provide information about the optimal posology of rhGH for each patient in order, therefore, to predict its adverse events and efficacy.

In addition, it has been shown that the effects mediated by the somatotropic hormone on some tissues are direct, therefore independent of the action of IGF1, whose plasma levels are not, in this case, predictive of therapeutic response.

For this reason, it is therefore necessary to identify a more specific biomarker capable of monitoring the efficacy, individual responsiveness and any adverse events in patients receiving somatotropic hormone.

The GH receptor (GHR) is expressed in several cells, including monocytes. It is therefore possible that the response of monocytes to the somatotropic hormone partially mirrors that of the chondrocyte and other cell types. Given the difficulty of obtaining osteomuscular biopsies or specific body areas in which GH mediates its biological action, the published works have identified the specific cell line in which to study the molecular effects of the hormone in monocytes, thanks to their easy accessibility and high number of GHR.

In consideration of this, the investigators propose to stimulate monocytes of healthy and GHD children in vitro with rhGH and through next generation sequencing to identify the characteristic gene expression profile. The GH responsive genes identified with this study can be used for correlation studies on the response to rhGH treatment.

ELIGIBILITY:
Inclusion Criteria:

* Height lower the 3th percentile

Exclusion Criteria:

* Any endocrinopathy
* Liver, kidney or haemolymphopoietic system disorders
* Celiac disease or other chronic malabsorption conditions
* Genetic syndromes (such as Turner's S., Cystic fibrosis or Down S.)
* Drug therapies interfering with growth

Ages: 6 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
gene expression in monocytes of GHD children | one year
  analysis of RNA-seq of monocytes of healthy and GHD children

SECONDARY OUTCOMES:
gene expression in monocytes modulated by GH | one year
  analysis of RNA-seq of monocytes of healthy and GHD children, stimulated with GH in culture

CONTACTS AND LOCATIONS:
Overall Officials: Mario Vitale, MD, Study Director — University of Salerno
Locations (1):
- Department of Medicine and Surgery, Univeristy of Salerno, Baronissi, Salerno, Italy

IPD SHARING:
Plan to Share IPD: Undecided